CLINICAL TRIAL: NCT05758883
Title: Post-approval Follow-up Study of the IC-8 Apthera IOL
Brief Title: Post-approval Follow-up Study of the IC-8 Apthera Intraocular Lens (IOL)
Status: Completed | Type: Observational
Sponsor: AcuFocus, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAIL-101-PAS
Record Dates: First submitted 2023-02-02; First posted 2023-03-08 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IC-8 Apthera intraocular lens (IOL) Group: Patients previously enrolled in the IC-8 Apthera IOL Investigational Device Exemption (IDE) study (G180075) and implanted with the IC-8 Apthera IOL.

SUMMARY:
The purpose of this study is to evaluate the long-term safety of the IC-8 Apthera intraocular lens (IOL).

DETAILED DESCRIPTION:
A prospective, multi-center, open-label, single-group, post-approval follow-up study of IC-8 Apthera intraocular lens (IOL) subjects previously implanted with the IC-8 Apthera IOL in the Investigational Device Exemption (IDE) clinical study (G180075). All subjects will undergo one scheduled study visit, which is the 3-year post IC-8 Apthera IOL implantation visit. There is one study group: subjects enrolled in the US IDE study (G180075) and implanted with the IC-8 Apthera IOL.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Investigational Device Exemption (IDE) G180075 study and implanted with the IC-8 Apthera intraocular lens (IOL)
* Able to comprehend and have signed a statement of informed consent
* Availability, willingness, ability and sufficient cognitive awareness to comply with examination procedures and study visit(s)

Exclusion Criteria:

* There are no exclusion criteria for this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential study subjects will be recruited from patients previously enrolled in the IC-8 Apthera intraocular lens (IOL) Investigational Device Exemption (IDE) study (G180075) and implanted with the IC-8 Apthera IOL.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Rates of secondary surgical interventions (SSIs) | 3 years post IC-8 Apthera IOL implantation
  Rates of secondary surgical interventions in the IC-8 Apthera intraocular lens (IOL) eyes will be assessed from the time the patient exited United States Investigational Device Exemption (IDE) G180075 through the Study visit
Rates of other serious adverse events | 3 years post IC-8 Apthera IOL implantation
  Rates of other serious adverse events in the IC-8 Apthera intraocular lens (IOL) eyes will be assessed from the time the patient exited United States Investigational Device Exemption (IDE) G180075 through the Study visit
Rates of ocular adverse events | 3 years post IC-8 Apthera IOL implantation
  Rates of ocular adverse events in the IC-8 Apthera intraocular lens (IOL) eyes will be assessed from the time the patient exited United States Investigational Device Exemption (IDE) G180075 through the Study visit
Rates of subjective visual disturbances | 3 years post IC-8 Apthera IOL implantation
  Rates of subjective visual disturbances will be assessed using responses to patient Reported Outcomes (PRO) and responses to non-directed question(s)

OTHER OUTCOMES:
Monocular best-corrected distance visual acuity (BCDVA) in IC-8 Apthera eyes and fellow eyes | 3 years post IC-8 Apthera IOL implantation
  Monocular best-corrected distance visual acuity will be assessed at the Study visit in the IC-8 Apthera intraocular lens (IOL) eyes and in the fellow eyes
Rate of intraocular lens (IOL) removals due to visual/optical reasons in the IC-8 Apthera eyes and fellow eyes | 3 years post IC-8 Apthera IOL implantation
  Rate of intraocular lens (IOL) removals (based on eyes with events) will be assessed at the Study visit in the IC-8 Apthera IOL eyes and in the fellow eyes
Mean monocular uncorrected distance visual acuity (UCDVA), uncorrected intermediate visual acuity (UCIVA) and uncorrected near visual acuity (UCNVA) | 3 years post IC-8 Apthera IOL implantation
  Mean monocular uncorrected distance visual acuity (UCDVA), uncorrected intermediate visual acuity (UCIVA) and uncorrected near visual acuity (UCNVA) will be evaluated in the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes
Mean distance-corrected intermediate visual acuity (DCIVA) and distance-corrected near visual acuity (DCNVA) | 3 years post IC-8 Apthera IOL implantation
  Mean distance-corrected intermediate visual acuity (DCIVA) and distance-corrected near visual acuity (DCNVA) will be evaluated in the IC-8 Apthera intraocular lens (IOL) eyes and the fellow eyes
Uncorrected distance visual acuity (UCDVA), uncorrected intermediate visual acuity (UCIVA), uncorrected near visual acuity (UCNVA) in IC-8 Apthera eyes and the fellow eyes in postoperative Manifest Refraction Spherical Equivalent (MRSE) groups | 3 years post IC-8 Apthera IOL implantation
  Uncorrected distance visual acuity (UCDVA), uncorrected intermediate visual acuity (UCIVA), uncorrected near visual acuity (UCNVA) in IC-8 Apthera eyes and the fellow eyes may be evaluated in postoperative Manifest Refraction Spherical Equivalent groups: -1.01 D to more myopic, -1.00 D to -0.50 D, -0.49 D to -0.25 D, -0.24 D to 0.00 D, +0.01 D to +0.25 D, +0.26 D to more hyperopic.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Fishkind, Bakewell, Maltzman, Hunter & Associates Eye Care & Surgery Center, Tucson, Arizona
  - Empire Eye & Laser Center, Bakersfield, California
  - Harvard Eye Associates, Laguna Hills, California
  - Altos Eye Physicians, Los Altos, California
  - Advanced Vision Care, Los Angeles, California
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Chu Vision Institute, Bloomington, Minnesota
  - Pepose Vision Institute, St Louis, Missouri
  - Kugler Vision, Omaha, Nebraska
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - Physicians Protocol, Greensboro, North Carolina
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - Bucci Laser Vision, Wilkes-Barre, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Baylor College of Medicine, Houston, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Hoopes Vision, Draper, Utah
  - Utah Eye Centers, Ogden, Utah
  - Virginia Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No